CLINICAL TRIAL: NCT02362360
Title: Investigation of a New 2-piece Ostomy Product in People With an Ileostomy or Colostomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: CP255
Record Dates: First submitted 2015-02-09; First posted 2015-02-12 (Estimated); Results first posted 2016-10-11 (Estimated); Last update posted 2016-10-11 (Estimated); Status verified 2016-08

CONDITIONS: Ileostomy; Colostomy
Keywords: Ostomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Coloplast Test Product then Comparator (Experimental): The subject first tests the Coloplast Test Product and then tests the Comparator
  Interventions: Device: Coloplast Test Product; Device: Comparator (Hollister)
- Comparator then Coloplast Test Product (Experimental): The subject first tests the Comparator and then tests the Coloplast Test Product.
  Interventions: Device: Coloplast Test Product; Device: Comparator (Hollister)

INTERVENTIONS:
Device: Coloplast Test Product — A new 2-piece ostomy appliance developed by Coloplast A/S
Device: Comparator (Hollister) — Comparator is a Hollister FlexWear baseplate (ileostomy) or a Hollister SoftFlex baseplate (colostomy) both used with a Hollister open bag.

SUMMARY:
The purpose of this study is to investigate the influence of a new ostomy product on the peristomal fit for people with an ileo- or colostomy.

ELIGIBILITY:
Inclusion Criteria:

* Have given written informed consent and in DK: signed a letter of authority
* Be at least 18 years of age and have full legal capacity
* Have had their ileostomy or colostomy for at least 3 months
* Able to use a baseplate size 15 to 40 mm
* Be able to handle the product themselves
* Normally experience faeces under the baseplate at least 3 times during 2 weeks
* Currently using a 2-piece flat product with mechanical coupling
* Willing to test both the Coloplast test product and the comparator product
* Willing to use an open bag size maxi during the investigation
* Willing to use Coloplast test product and comparator products without initial use of accessories (except tube paste / belt)
* Willing to use at least 1 baseplate every 3rd day during the investigation
* Is able to use a custom cut product
* Be suitable for participating in the investigation

Exclusion Criteria:

* Are currently receiving or have within the past 2 months received radio-and/or chemotherapy (low doses chemotherapy are allowed for other indications than cancer)
* Are currently receiving or have within the past month received topical steroid treatment in the peristomal skin area (lotion or spray). Systemic steroid (tablet/injection) treatment are allowed
* Are pregnant or breastfeeding
* Are participating in other interventional clinical investigations or have previously participated in this investigation
* Use irrigation during the investigation (flush the intestines with water)
* Are currently suffering from peristomal skin problems i.e. bleeding and/or broken skin (assessed by the investigator)
* Have a loop ostomy
* Have known hypersensitivity towards any of the products used in the investigation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2015-02; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- Trial Form Support ApS (TFS), Soeborg, Denmark
- Germany (2):
  - Charité - Universitätsmedizin Berlin, Klinik für Allgemein-, Gefäß- und Thoraxchirurgie, Berlin
  - SIEWA Coloplast Homecare, Hamburg
- QPS Netherlands, Groningen, Netherlands
- Sykepleierklinikken A/S, Larvik, Larvik, Norway

REFERENCES:
- [Derived] Rolfsen T, Vestergaard M, Hansen MF, Boisen EB, Dambaek MR. Body Fit With a Pouching System With Concave Contour for People With an Outward Peristomal Body Profile: Effects on Leakage, Wear Time, and Quality of Life: A Randomized Controlled Cross-Over Trial. J Wound Ostomy Continence Nurs. 2024 Jul-Aug 01;51(4):303-311. doi: 10.1097/WON.0000000000001088. Epub 2024 Jul 19. PMID 39037163

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One subject was a screen failure and was not exposed to any of the test products. This subject was excluded from the safety population, which therefore included 52 subjects.
Period: Period 1
Arm/Group | Coloplast Test Product Then Comparator | Comparator Then Coloplast Test Product
Started | 26 | 26
Completed | 23 | 25
Not Completed | 3 | 1
Not completed — Lack of Efficacy | 1 | 0
Not completed — Withdrawal by Subject | 2 | 1
Period: Period 2
Arm/Group | Coloplast Test Product Then Comparator | Comparator Then Coloplast Test Product
Started | 23 | 25
Completed | 23 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Study Population: All subjects included in the investigation
Arm/Group | Overall Study Population
Number analyzed (Participants) | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.9 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 41

OUTCOME MEASURES:

1. Primary Outcome: Fit to the Peristomal Area, Measured by a 5-point Scale Ranging From "Very Poor" to "Very Good".
Description: Subjects will evaluate the fit to body for each product by answering the question "How was the baseplates ability to fit to the body contours in the area around the stoma?". The question is answered with a 5-point scale ranging from "very poor" to "very good".
Time Frame: 21 +/- 3 days
Measure: Number; unit: percentage of subjects answering
Groups:
- Coloplast Test Product: Answers from subjects testing Coloplast test product
- Comparator: Answers from subjects testing Comparator
Arm/Group | Coloplast Test Product | Comparator
Number analyzed (Participants) | 51 | 49
percentage of subjects answering
  Very good | 56.9 | 10.6
  Good | 29.4 | 27.7
  Acceptable | 9.8 | 42.6
  Poor | 3.9 | 19.1
  Very poor | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the study period: 42 days +/- 6 days
Arm/Group | Coloplast Test Product | Comparator
Serious Adverse Events (participants affected / at risk) | 0/51 | 3/49
Other Adverse Events (participants affected / at risk) | 9/51 | 17/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Coloplast Test Product (N=51) | Comparator (N=49)
Lung infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — not related to Comparator product
Compartment syndrome in left lower leg (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — not related to Comparator product
Acute renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) — not related to Comparator product
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Coloplast Test Product (N=51) | Comparator (N=49)
Skin irritation (Skin and subcutaneous tissue disorders) | 9 (14) | 17 (21) — related adverse events to either Test product or Comparator (adverse event categorised as unlikely related, probably related, possibly related and definitly related are treated as related adverse events).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less